CLINICAL TRIAL: NCT05019248
Title: A Non-interventional Observation Study to Evaluate Immune Responses Following Seasonal Influenza Vaccine in Participants With Relapsing Multiple Sclerosis Treated With Cladribine Tablets
Brief Title: Immune Response to Seasonal Influenza Vaccination in Multiple Sclerosis Patients Receiving Cladribine
Acronym: CIRMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1474
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Vaccine Response Impaired
Keywords: influenza vaccination; cladribine
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — (I) Serum samples for assessment of antibody levels (II) Peripheral blood mononuclear cells for assessment of cellular immune responses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- vaccination prior to first cladribine exposition
  Interventions: Biological: Most recent vaccine to seasonal influenza
- vaccination shortly after first cladribine exposition
  Interventions: Biological: Most recent vaccine to seasonal influenza
- vaccination prior to second cladribine exposition
  Interventions: Biological: Most recent vaccine to seasonal influenza
- vaccination following completion of cladribine treatment
  Interventions: Biological: Most recent vaccine to seasonal influenza
- vaccination in patients with RRMS not subjected to cladribine
  Interventions: Biological: Most recent vaccine to seasonal influenza

INTERVENTIONS:
Biological: Most recent vaccine to seasonal influenza — Seasonal Influenza vaccine: according to the latest SmPC and according to national guidelines (published by the Standing Committee on Vaccination (STIKO)).

SUMMARY:
The primary objective of this study is to characterize the antibody response to seasonal influenza vaccine, in patients with active RRMS, treated with cladribine, compared to control individuals with basic immunomodulatory treatment. Serum antibody titers against the respective pathogen will be assessed prior to and 6 to 8 months following vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF)
2. Age 18 to 60 years old (inclusive) as of the date the ICF is signed
3. Diagnosis of RRMS according to the revised McDonald criteria
4. EDSS score of 0.0 to 7.0 (inclusive)
5. In case of participants who are subjected to influenza vaccination by the treating physicians prior to cladribine the first or second cycle of cladribine (cohort 1 + cohort 3), this should be performed at least 4 to 6 weeks before the start of cladribine.

Definition of control group:

Patients with active RRMS treated with cladribine will be compared to sex and age matched control individuals, with RRMS under basic treatment either with interferon beta, glatiramer acetate, dimethyl fumarate or teriflunomide, who provide sample material prior to and 6 to 8 months after routine seasonal influenza vaccination during the same period.

Exclusion Criteria:

1. Previous treatment with B-cell targeted therapies (e.g., rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab)
2. Any previous treatment with alemtuzumab, cladribine, cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, or bone marrow transplantation
3. Medical, psychiatric, cognitive, or other conditions that, in the investigator's opinion, compromise the patient's ability to understand the patient information, to give informed consent, or to complete the study
4. Patients that receive immunosuppressive treatment for diseases other than MS or that receive long-term corticosteroid treatment
5. Patients that received apheresis procedures 6 weeks prior to vaccination or in-between vaccination and DMT initiation
6. Systemic high dose corticosteroid therapy within 6 weeks prior to vaccination or in-between vaccination and DMT initiation
7. Patients with verified infection by human-immunodeficiency-virus or hepatitis-c-virus
8. Patients with major impairment of the blood coagulation system including therapy with anticoagulants
9. Patients with known chicken egg allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 52 patients per group/cohort, resulting in a theoretical maximum number of 260 patients. Patients will be screened until this number is reached.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion who achieve seroprotection | 6 months
  The capacity of influenza vaccine to elicit a measurable immune response (immunogenicity) when it is administered (i) shortly (at least 4-6 weeks) before cladribine initiation (cohort 1), (ii) 3 to 4 months after cladribine initiation (cohort 2) (iii) shortly (at least 4-6 weeks) before second cladribine administration (cohort 3) and (iv) in patients who have already received the second cycle of cladribine tablets (3 to 4 months after second cycle; cohort 4), compared to RRMS patients treated with basic DMTs (cohort 5). Efficacy is measured as proportion of patients who achieve seroprotection (specific hemagglutination inhibition (HI) titers > 1:40)).

SECONDARY OUTCOMES:
Fraction with 2-fold increase of HI titers | 6 months
  Proportion of patients who achieve a 2-fold increase in specific HI titers at 6 to 8 months post-immunization
Fraction with 4-fold increase of HI titers | 6 months
  Proportion of patients who achieve a 4-fold increase in specific HI titers at 6 months post-immunization
Seroconversion rate | 6 months
  Proportion of patients with seroconversion (i.e., a pre-vaccination antibody titer < 10 and a post-vaccination HI titer > 40)
Mean antibody titers | 6 months
  Geometric mean antibody titers (GMTs) and geometric mean antibody ratios (GMRs, post-vaccination:pre-vaccination) prior and 6 months after vaccination
Cellular immune responses | 6 months
  Flow cytometry analysis, which will include (but is not limited to) the following cells: Total B cells (CD19 positive), B-cell subsets, e.g., memory B cells, naïve B cells, plasma cells; Total T cell (CD3 positive) and T cell subsets, e.g. T helper cells, cytotoxic lymphocyte T cells
Serum immunoglobulin subtypes | 6 months
  Analysis of quantitative Ig levels (including total Ig, IgG, IgG subtypes, IgM, and IgA)
Influenza infections | 6 months
  Incidence of infections caused by influenza

CONTACTS AND LOCATIONS:
Overall Officials: Sven G Meuth, MD, PhD, Principal Investigator — Heinrich-Heine-University Duesseldorf, Germany
Locations (1):
- Medical Faculty, Heinrich-Heine-University, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rolfes L, Pfeuffer S, Skuljec J, He X, Su C, Oezalp SH, Pawlitzki M, Ruck T, Korsen M, Kleinschnitz K, Aslan D, Hagenacker T, Kleinschnitz C, Meuth SG, Pul R. Immune Response to Seasonal Influenza Vaccination in Multiple Sclerosis Patients Receiving Cladribine. Cells. 2023 Apr 25;12(9):1243. doi: 10.3390/cells12091243. PMID 37174643